CLINICAL TRIAL: NCT06252155
Title: The Effect of Music Played to Newborn Mothers on Postpartum Blues: Randomized Controlled Study
Brief Title: The Effect of Music Played to Newborn Mothers on Postpartum Blues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Burcu KUCUKKAYA, Asst. Prof, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023-03
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Postpartum Blues; Birth Depression; Mothers
Keywords: Music
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Before starting the research, two groups of mothers will be randomly formed. As a randomization method, mothers who meet the sampling inclusion criteria determined in the research will be identified and listed. Individuals to be taken into two groups will be determined by randomization method from the random numbers table. (http://www.stattrek.com/statistics/randomnumber-generator.aspx).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No intervention will be made to the control group.
- Music Group (Experimental): Mothers will listen to music for 30 minutes every day for 2 postpartum days. The type of music to be used in this study will be Turkish music . Turkish music will be preferred in the study because it is a part of the culture in which the study will be conducted. This type of music was preferred because it evokes feelings of happiness, laughter, joy, power, courage and heroism in the human soul. In deciding the type of music listened to in the study, expert opinion was taken from a faculty member teaching music therapy at a state university. During the music session, the mother will take a comfortable position on the sofa or bed. She will also be asked to close her eyes and imagine where she wants to be. She will also be asked to breathe slowly and deeply to regulate her breathing.
  Interventions: Other: Music

INTERVENTIONS:
Other: Music — Mothers will listen to music for 30 minutes every day for 2 postpartum days. The type of music to be used in this study will be Turkish music . Turkish music will be preferred in the study because it is a part of the culture in which the study will be conducted. This type of music was preferred because it evokes feelings of happiness, laughter, joy, power, courage and heroism in the human soul. In deciding the type of music listened to in the study, expert opinion was taken from a faculty member teaching music therapy at a state university. During the music session, the mother will take a comfortable position on the sofa or bed. She will also be asked to close her eyes and imagine where she wants to be. She will also be asked to breathe slowly and deeply to regulate her breathing. The mother will be told to feel comfortable, to feel her body relax from head to toe while listening to music, to focus on the music and to free her thoughts.
  Arms: Music Group

SUMMARY:
The prospective and two-arm randomized controlled study was conducted on n = 82 (41 = control, 41 = music group) mothers who gave birth at term at Trakya University Health Research and Application Center Maternity Service between May and December 2023. The music group was listened to Turkish music played for 30 minutes every day for 2 postpartum days. Research data were collected through the "Personal Information Form", "Stein Blues Scale (SDS)" and Edinburgh Postpartum Depression Scale (EPDS). The scales used in the research were evaluated four times: pre-, intermediate, follow-up and post-test. Descriptive statistics, Pearson and Spearman's correlation analyzes will be used in the analysis of research data.

DETAILED DESCRIPTION:
Type of Research This study was conducted in a prospective, two-arm and randomized controlled manner.

Where the Research Was Conducted The research was conducted on mothers who gave birth at Trakya University Health Research and Application Center Maternity Service between May and December 2023.

Population/Sample of the Research The power analysis of the study was performed with the G*POWER 3.1.9.7 (Power analysis statistical software) program. To determine the sample size of the study, to measure the effect of music applied to mothers with term babies on postpartum blues, 41 control groups and 41 control groups were used to test a difference in the predicted medium effect size (d=.5) based on our clinical observation with a 5% margin of error and 80% power value. It was calculated that a total of 82 mothers, 41 in the intervention group, should be included in the study.

Data Collection Tools-Validity and Reliability Information In the study, "Personal Information Form", "Stein Blues Scale" and "Edinburgh Postpartum Depression Scale", which were created by the researchers by scanning the literature, were used.

Personal Information Form: Containing the personal characteristics of mothers who have just given birth (age, mother's education level, mother's employment status, family type, spouse's age, spouse's education status, spouse's employment status, income status, place of residence, smoking status, alcohol use status, 12 questions regarding physical exercise status, 10 questions about obstetric characteristics (number of pregnancies, number of live births, number of children, number of miscarriages, number of curettages, type of birth, intentional pregnancy status, planned pregnancy status, gender of the baby, week of birth of the baby), psycho-social characteristics (the state and frequency of feeling tense in daily life, the methods used to calm down when tense in daily life, the situation of using traditional and complementary methods to calm down when tense in daily life, and which method is used to calm down when tense in daily life, the traditional and complementary methods used to calm down when tense in daily life). If using complementary methods, sharing with the source of information and healthcare personnel, current emotional state, emotional state regarding pregnancy, psychological support from spouse during pregnancy, psychological support from relatives (such as mother/sibling) during pregnancy, social status during pregnancy. It consists of a total of 34 questions, 12 of which are evaluating relationships, spending time with friends during pregnancy.

Stein Blues Scale (SBS): Stein used this scale for the first time in a study in which 37 women were included in the first postpartum week and then followed for 3 months. The scale consists of two parts with a total of 13 questions. The first 8 questions are likert-type questions that examine mood symptoms. In the second part, the answers are yes/no; There are 5 questions investigating the presence of symptoms such as headache, restlessness, difficulty concentrating, forgetfulness and confusion. While the scoring of the section containing Likert-type questions varies between 0-4, if there is a symptom in the last 5 questions, 1 point for each is added to the total score. The minimum score is 0 while the maximum score is 26. Patients are asked to answer the scale thinking only of that day. While mild blues symptoms apply to scores between 3 and 8, scores of 8 and above indicate severe blues symptoms. Stein tested the validity and reliability of the scale according to the 60-question self-administered Goldberg Scale (r = .80) and found its reliability to be r = .70. Stein scale questions screen for symptoms of depression, crying, restlessness, anxiety, fatigue, tension, irritability, poor concentration, forgetfulness, confusion, anorexia, daydreaming and headache in women who have just given birth. In this study, the Cronbach's Alpha value of the scale was determined as .99.

Edinburgh Postpartum Depression Scale (EPDS); to determine the risk of depression in women in the postpartum period. EPDS is used in our country and the Cronbach Alpha value of the scale was found to be .87. The answers to the 4-point Likert type scale consisting of 10 questions are scored between 0-3. The cut-off score for the scale was taken as 12/13. If the score obtained is 12 and below, the patient is considered not at risk for postpartum depression, and if it is 13 and above, the patient is considered at risk for postpartum depression. Scores from the scale range from 0 to 30.

Procedure Mothers who met the inclusion criteria of the study were visited in the maternity ward within the first 12 hours after birth and offered to participate in the study. Participants were given a consent form containing information stating that previous studies had shown the positive effects of singing on various aspects of well-being and that the intervention was therefore designed to investigate the effects of listening to music on emotional changes in the postnatal context. After obtaining informed written consent, they were randomized to the control or intervention group and received the baseline questionnaire, which included the "Personal Information Form", the "Stein Blues Scale" and the "Edinburgh Postpartum Depression Scale". A member of the study team went to the ward where the study was conducted for 2 days to collect the completed questionnaire, and when he went to collect the completed questionnaire for the last time, he gave the mothers a small gift as a thank you for their participation in the study. After the initial measurement, the mother was asked to listen to the selected music within 12 hours and repeat the scales after listening to the music. 24 hours after the first music listening application, the mother was asked to apply the same scales again, listen to the music, and repeat the scales as the final test. An overview of the procedure. Information about the flow and which survey was administered when is given.

Music application: Mothers will listen to music for 30 minutes every day for 2 postpartum days. The type of music to be used in this study will be Turkish music works played . Turkish music will be preferred in the study because it is a part of the culture in which the study will be conducted. This type of music was preferred because it evokes feelings of happiness, laughter, joy, power, courage and heroism in the human soul . In deciding the type of music listened to in the study, expert opinion was taken from a faculty member teaching music therapy at a state university. During the music session, the mother will take a comfortable position on the sofa or bed. She will also be asked to close her eyes and imagine where she wants to be. She will also be asked to breathe slowly and deeply to regulate her breathing. The mother will be told to feel comfortable, to feel her body relax from head to toe while listening to music, to focus on the music and to free her thoughts. The mother will start listening to the piece with the help of the researchers' phone and a portable Bluetooth speaker, wireless sound bomb, or headphones. The volume of the music will be set at 60-66 beats per minute .

Ethical Aspect of Research For the ethical suitability of the research, the Istanbul Kent University Health Sciences Scientific Research and Publication Ethics Board meeting dated 25.04.2023 and numbered 2023-03 received ethical approval and written permission from the Chief Physician of Trakya University Health Research and Application Center for the collection of data and a newborn who agreed to participate in the study. Written informed consent was obtained from the mothers who participated. The research was carried out in accordance with the rules of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-49,
* To can read, understand and write Turkish,
* Had a term birth (single birth at 38 weeks and above),
* Had a normal vaginal delivery or cesarean delivery after an uncomplicated pregnancy,
* Has stable vital signs, who is undergoing infertility treatment not having any chronic disease (such as hypertension, diabetes mellitus),
* Do not experiencing serious depression, anxiety and stress, not having any organic or non-organic disease that may cause cognitive impairment (such as delirium, dementia, mental retardation, etc.),
* Not having serious maternal complications,
* Mothers who volunteered to participate in the study

Exclusion Criteria:

* Under 18 and over 49 years of age,
* Preterm birth (under 37 weeks and/or multiple birth),
* After a complicated pregnancy, birth has not been completed by normal vaginal delivery or cesarean delivery method,
* Without stable vital signs,
* Those who have received infertility treatment,
* Having a chronic disease (such as hypertension, diabetes mellitus),
* Experiencing serious depression, anxiety and stress,
* Having any organic or non-organic disease that may cause cognitive impairment (such as Delirium, Dementia, Mental Retardation, etc.),
* Serious maternal complications,
* Mothers who did not volunteer to participate in the research

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 82 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Postpartum blues evaluated using the Edinburgh Postpartum Depression Scale | change from baseline and 1 and 2 day of practice.
  It was created by George S. Stein in 1980. Stein used this scale for the first time in a study in which 37 women were included in the first postpartum week and then followed for 3 months. The scale consists of two parts with a total of 13 questions. The first 8 questions are likert-type questions that examine mood symptoms. In the second part, the answers are yes/no; There are 5 questions investigating the presence of symptoms such as headache, restlessness, difficulty concentrating, forgetfulness and confusion. While the scoring of the section containing Likert-type questions varies between 0-4, if there is a symptom in the last 5 questions, 1 point for each is added to the total score. The minimum score is 0 while the maximum score is 26. Patients are asked to answer the scale thinking only of that day (23). While mild blues symptoms apply to scores between 3 and 8, scores of 8 and above indicate severe blues symptoms.
Depression evaluated using the Stein Blues Scale | change from baseline and 1 and 2 day of practice.
  Cox et al. (1987) to determine the risk of depression in women in the postpartum period. EPDS is used . The answers to the 4-point Likert type scale consisting of 10 questions are scored between 0-3. The cut-off score for the scale was taken as 12/13. If the score obtained is 12 and below, the patient is considered not at risk for postpartum depression, and if it is 13 and above, the patient is considered at risk for postpartum depression. Scores from the scale range from 0 to 30.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Bartın, Turkey (Türkiye)

REFERENCES:
- [Derived] Kucukkaya B, Can I, Guler G. The effect of music played to new birth mothers on postpartum blues: A randomized controlled trial. Early Hum Dev. 2024 May;192:106013. doi: 10.1016/j.earlhumdev.2024.106013. Epub 2024 Apr 17. PMID 38657398